CLINICAL TRIAL: NCT03338998
Title: A Phase II, Patient- and Investigator-blinded, Randomized, Placebo-controlled Study to Evaluate Efficacy, Safety and Tolerability of BAF312 (Siponimod) in Patients With Stroke Due to Intracerebral Hemorrhage (ICH)
Brief Title: Efficacy, Safety and Tolerability of BAF312 Compared to Placebo in Patients With Intracerebral Hemorrhage (ICH).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CBAF312X2207
Record Dates: First submitted 2017-11-08; First posted 2017-11-09 (Actual); Results first posted 2021-06-07 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Hemorrhagic Stroke; Intracerebral Hemorrhage (ICH)
Keywords: stroke; intracerebral hemorrhage; ICH; BAF312; siponimod; sphingosine-1-phosphate receptor; adult
MeSH Terms: conditions — Hemorrhagic Stroke; Cerebral Hemorrhage; Stroke | interventions — siponimod

STUDY DESIGN:
Intervention Model Description: This is a randomized, patient- and investigator-blinded, placebo-controlled, parallel group study of BAF312 on top of standard-of-care for ICH, consisting of 3 epochs: Screening/Baseline, Treatment (Day 1-14), and Follow-Up (to Day 90)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BAF312 (Experimental): Days 1 - 7, IV up titration; days 8 - 14, 10 mg (5 x 2 mg tablets) taken daily orally
  Interventions: Drug: BAF312 solution; Drug: BAF312 tablet
- Placebo (Placebo Comparator): Days 1 - 7, IV up titration; days 8 - 14, 10 mg (5 x 2 mg tablets) taken daily orally - matching placebo
  Interventions: Drug: Matching Placebo for BAF312 solution; Drug: Matching Placebo for BAF312 tablet

INTERVENTIONS:
Drug: BAF312 solution — Solution for intravenous (IV) infusion - 4.5mg/4.5mL
  Other Names: Siponimod
  Arms: BAF312
Drug: Matching Placebo for BAF312 solution — Solution for intravenous (IV) infusion - 0mg/4.5mL matching placebo
  Arms: Placebo
Drug: BAF312 tablet — 2 mg film-coated tablet
  Other Names: Siponimod
  Arms: BAF312
Drug: Matching Placebo for BAF312 tablet — 0 mg film-coated tablet matching placebo
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled, subject and investigator-blinded study to evaluate efficacy, safety and tolerability of BAF312 in participants with intracerebral hemorrhage (ICH)

DETAILED DESCRIPTION:
This was the first trial of BAF312 in ICH patients to evaluate if BAF312 had the potential to limit brain inflammation after ICH, and thereby improve neurological outcome for stroke patients when administered in addition to standard of care.

ICH patients meeting study criteria were randomized at 1:1 ratio into either active or placebo group. Patients received an intravenous infusion (i.v.) treatment within 24 hours of an ICH event and were up titrated for 7 days. Following the i.v. treatment, participants received 10 mg BAF312 or placebo in tablet form (taken daily orally) for an additional 7 days. Participants were followed for an additional 76 days after treatment for neurological and safety conditions during three clinic visits.

Recruitment for the trial was put on hold due to the COVID-19 pandemic. Thirty-two patients had been enrolled in the trial and completed the protocol as planned. After seven months of the trial being on hold, an Interim analysis was conducted and reviewed by the Data Monitoring Committee. Novartis terminated the trial due to lack of potential efficacy.

ELIGIBILITY:
Inclusion Criteria:

ICH patients eligible for inclusion in this study must fulfill all of the following criteria:

1. Male or female patients aged 18 to 85 years (inclusive).
2. Written informed consent obtained before any study assessment is performed. If the patient is not able to give the informed consent personally, consent by a relative or legal representative is acceptable.
3. Spontaneous, supratentorial intracerebral hemorrhage in cerebral cortex or deep brain structures (putamen, thalamus, caudate, and associated deep white matter tracts) with a volume ≥ 10 mL but ≤ 60 mL (calculated by the ABC/2 method, after Kothari et al 1996) determined by routine clinical MRI or CT.
4. Patients with the onset of ICH witnessed and/or last seen healthy no longer than 24 hrs previously.
5. Patients with Glasgow Coma Scale (GCS) best motor score no less than 5 (brings hands above clavicle on stimulus to head or neck).

Exclusion Criteria:

ICH patients fulfilling any of the following criteria are not eligible for inclusion in this study:

1. Use of other investigational drugs within 5 half-lives of enrollment, or until the expected pharmacodynamic effect has returned to baseline (for biologics), whichever is longer.
2. History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes (e.g., fingolimod).
3. Current use of concomitant medications with potent CYP2C9/3A4 inhibitory or induction potential.
4. Infratentorial (midbrain, pons, medulla, or cerebellum) ICH.
5. Candidates for surgical hematoma evacuation or other urgent surgical intervention (i.e., surgical relief of increased intracranial pressure) on initial presentation. If during the treatment period surgical hematoma evacuation or surgical intervention to lower intracranial pressure becomes indicated, the investigational treatment should be stopped.
6. Patients with intraventricular hemorrhage (IVH) having a Graeb score of >3 on initial presentation. Patients must not have blood in the 4th ventricle and may only have blood in the 3rd ventricle in the absence of ventricular expansion. Trace or mild hemorrhage in either or both lateral ventricles is permitted. Patients with hydrocephalus determined radiologically on initial presentation are excluded regardless of Graeb score.
7. Secondary ICH due to:

   * aneurysm
   * brain tumor
   * arteriovenous malformation
   * thrombocytopenia, defined as platelet count of <150,000/µl
   * known history of coagulopathy
   * acute sepsis
   * traumatic brain injury (TBI)
   * disseminated intravascular coagulation (DIC)
8. Prior disability due to other disease compromising mRS evaluation, thereby interfering with the primary outcome, operationally defined as an estimated mRS score (by history) of ≥ 3 before ICH for patients less than or equal to 80 years of age. For ICH patients 81-85 years of age, estimated mRS by history prior to ICH must be less than or equal to 1 (no significant disability despite symptoms).
9. Preexisting unstable epilepsy.
10. Patients with active systemic bacterial, viral or fungal infections.
11. Concomitant drug-related exclusion criteria:

    * Intravenous immunoglobulin, immunosuppressive and/or chemotherapeutic medications.
    * Moderate immunosuppressives (e.g. azathioprine, methotrexate) and/or fingolimod within 2 months prior to randomization.
    * Stronger immunosuppressives (e.g. cyclophosphamide, immunosuppressive mAb) within (minimally) 6 months prior to randomization, or longer with long-lasting immunosuppressive medications as determined by the investigator.
12. Cardiovascular exclusion criteria:

    * Cardiac conduction or rhythm disorders including sinus arrest or sino-atrial block, heart rate <50 bpm, sick-sinus syndrome, Mobitz Type II second degree AV block or higher grade AV block, or preexisting atrial fibrillation (either by history or observed at screening).
    * PR interval >220 msec. Long QT syndrome or QTcF prolongation >450 msec in males or >470 msec in females on screening electrocardiogram (ECG).
    * Patients receiving treatment with QT-prolonging drugs having a long half-life (e.g., amiodarone).
13. Any of the following abnormal laboratory values prior to randomization:

    * White blood cell (WBC) count < 2,000/μl (< 2.0 x 109/L)
    * Lymphocyte count < 800/μl (< 0.8 x 109/L)
14. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
15. Patients with any other medically unstable condition or serious laboratory abnormality as determined by the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-12-24 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2020-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin N. Sheth, MD, Principal Investigator — Yale University
Locations (10):
- United States (10):
  - Novartis Investigative Site, Palo Alto, California
  - Novartis Investigative Site, New Haven, Connecticut
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1084

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period
Arm/Group | BAF312 | Placebo
Started | 16 | 13
Completed | 8 | 10
Not Completed | 8 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 0 | 2
Not completed — Protocol deviation | 1 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Subject failed swallow test | 4 | 0
Period: Safety Follow-Up Period
Arm/Group | BAF312 | Placebo
Started | 16 | 13
Completed | 14 | 12
Not Completed | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Protocol deviation | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BAF312 | Placebo | Total
Number analyzed (Participants) | 16 | 13 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (13.6) | 63.8 (9.06) | 60.8 (11.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 6 | 7 | 13
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 8 | 11 | 19
  Black | 5 | 0 | 5
  Asian | 0 | 1 | 1
  Other | 3 | 1 | 4
Absolute perihematoma edema (aPHE) volume [Mean (Standard Deviation); unit: mL] | 32.927 (32.3153) | 22.825 (9.8617) | 28.237 (24.7188)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Perihematoma Edema (aPHE) Volume Measured by Computed Tomography (CT) Scan After Intracerebral Hemorrhage (ICH)
Description: Following the initial diagnostic CT, repeat CT images were obtained between 24-48 h after the diagnostic scan, and on Day 7 and Day 14 to capture the trajectory of PHE increase and plateau after ICH. Only non-contrast study CT scans were obtained on Day 7 and Day 14. The non-contrast scan acquired on each patient at first follow-up (i.e. 24-48 h after the diagnostic scan) served as the baseline for our analysis. All CT scans were uploaded through a secure server, and edema and hematoma volumes were measured in a semi-automated manner by one Central Reader.
Time Frame: On Day 14 following ICH
Population: Per protocol analysis set
Measure: Geometric Mean (90% Confidence Interval); unit: mL
Arm/Group | BAF312 | Placebo
Number analyzed (Participants) | 14 | 13
mL | 55.09 [42.444 to 71.509] | 52.50 [40.042 to 68.835]
Statistical Analysis 1: Comparison: BAF312 vs Placebo; Test type: Superiority; p = 0.585, ANCOVA; Geo-mean ratio = 1.05, 90% CI 2-sided [0.717 to 1.535]

2. Secondary Outcome: Plasma BAF312 Concentrations
Description: Blood samples will be collected to assess plasma concentrations.
Time Frame: Days 1, 8, and 14
Population: Pharmacokinetics analysis set that included participants with at least one blood sample available
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | BAF312
Number analyzed (Participants) | 11
ng/mL
  Day 1 - 0.1 Hours Post I.V. Dose n=11 | 0.1658 (85.6)
  Day 1 - 2 Hours Post I.V. Dose n=11 | 0.5663 (78.7)
  Day 1 - 6 Hours Post I.V. Dose n=10: number analyzed (Participants) | 10
  Day 1 - 6 Hours Post I.V. Dose n=10 | 2.4313 (30.5)
  Day 8 - 0 Hours Pre Oral Dose n=11 | 81.9423 (55.9)
  Day 14 - 0 Hours Pre Oral Dose n=11 | 36.4460 (550.8)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment (14 days) plus 76 days post treatment, up to approximately of 90 days
Groups:
- Total: Total
Arm/Group | BAF312 | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/13 | 0/29
Serious Adverse Events (participants affected / at risk) | 2/16 | 2/13 | 4/29
Other Adverse Events (participants affected / at risk) | 14/16 | 11/13 | 25/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BAF312 (N=16) | Placebo (N=13) | Total (N=29)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1
Septic shock (Infections and infestations) | 0 | 1 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Hypotension (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BAF312 (N=16) | Placebo (N=13) | Total (N=29)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 2
Bradycardia (Cardiac disorders) | 5 | 0 | 5
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 1
Dry eye (Eye disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 2 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2
Infusion site extravasation (General disorders) | 2 | 0 | 2
Infusion site irritation (General disorders) | 0 | 1 | 1
Injection site swelling (General disorders) | 1 | 0 | 1
Pain (General disorders) | 1 | 0 | 1
Peripheral swelling (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1
Swelling face (General disorders) | 0 | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Blood bicarbonate decreased (Investigations) | 1 | 0 | 1
Computerised tomogram abnormal (Investigations) | 0 | 1 | 1
Transaminases increased (Investigations) | 1 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1
Facial paralysis (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 2 | 3
Hydrocephalus (Nervous system disorders) | 1 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 2 | 2
Confusional state (Psychiatric disorders) | 1 | 0 | 1
Depression (Psychiatric disorders) | 2 | 0 | 2
Hallucination, visual (Psychiatric disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2 | 2
Restlessness (Psychiatric disorders) | 1 | 0 | 1
Sleep disorder (Psychiatric disorders) | 2 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1
Azotaemia (Renal and urinary disorders) | 1 | 1 | 2
Urinary retention (Renal and urinary disorders) | 1 | 2 | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/98/NCT03338998/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/98/NCT03338998/SAP_001.pdf